CLINICAL TRIAL: NCT06712849
Title: Multi-day Effect of Noninvasive Brain Stimulation in Adults With Amblyopia
Brief Title: Noninvasive Brain Stimulation in Adult Amblyopia
Acronym: NIBSAAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Arijit Chakraborty, Assistant Director of Research, Midwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRB-IL 23044
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Amblyopia
Keywords: Amblyopia; Non-invasive Brain Stimulation; Transcranial Random Noise Stimulation; Visual Perception; Visual Evoked Potentials
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham Stimulation (Sham Comparator): 40-minute sessions of sham stimulation for 5 consecutive days.
  Interventions: Device: Sham Transcranial Random Noise Stimulation
- hf-tRNS Stimulation (Active Comparator): 40-minute sessions of hf-tRNS stimulation for 5 consecutive days.
  Interventions: Device: High Frequency Transcranial Random Noise Stimulation

INTERVENTIONS:
Device: Sham Transcranial Random Noise Stimulation — Sham transcranial random noise stimulation will be applied over the primary visual cortex (area V1) with the current ramping up for 20 seconds before ramping down for 20 seconds. The 2.0 milliamp current stimulation will occur for only a few seconds at the start and at the end of the 40 minutes.
  Other Names: Sham tRNS
  Arms: Sham Stimulation
Device: High Frequency Transcranial Random Noise Stimulation — Non-invasive brain stimulation will involve the use of high-frequency transcranial random noise stimulation (100-640 Hz) to apply a 2.0 milliamp current over the primary visual cortex (area V1) for approximately 40 minutes with a ramp up to the maximum programmed current and ramp down of 20 seconds.
  Other Names: tRNS; hf-tRNS
  Arms: hf-tRNS Stimulation

SUMMARY:
The goal of this randomized controlled trial is to investigate the effectiveness of non-invasive brain stimulation in treating adults with amblyopia. The main questions it aims to answer are:

1. What are the effects of non-invasive brain stimulation on neuronal plasticity in the visual cortex of adults with amblyopia, and does it produce lasting changes?
2. Do cumulative sessions of non-invasive brain stimulation influence neural plasticity and higher-order visual functions in adults with amblyopia?

The investigators hypothesize that non-invasive brain stimulation will show a positive cumulative effect after five (5) consecutive days of stimulation on visual perception and function in adults with amblyopia.

Participants will be randomized into one of two treatment groups:

1. High-frequency transcranial random noise stimulation (hf-tRNS).
2. Sham stimulation.

Researchers will compare baseline measurements of crowded visual acuity, contrast sensitivity, stereoacuity, phosphene thresholds, global motion perception, form pattern recognition and pattern-reversal visual evoked potentials (VEPs) to post-treatment measurements for each group.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 55 years of age
* Formal diagnosis of amblyopia in one or both eyes of any etiology

Exclusion Criteria:

* History of optic nerve disease, including glaucoma and optic neuritis
* History of neurological conditions, including demyelinating disease or stroke
* Presence of metal or electronic implants in or on the body, including pacemakers
* Taking medications that can affect normal neurological function, including antipsychotics, antiepileptics, and opioids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Crowded Visual Acuity | Pre- and post-treatment (Days 1-5); 24-hour follow-up (Day 6); 72-hour follow-up (Day 8); and 10-day follow-up (Day 15).
  A change in crowded visual acuity is measured in LogMAR from baseline.
Stereo Acuity | Pre- and post-treatment (Days 1-5); 24-hour follow-up (Day 6); 72-hour follow-up (Day 8); and 10-day follow-up (Day 15).
  A change in stereo acuity is measured in arc seconds from baseline.
Phosphene Threshold | Pre- and post-treatment (Days 1-5); 24-hour follow-up (Day 6); 72-hour follow-up (Day 8); and 10-day follow-up (Day 15).
  A change in phosphene threshold (%) from baseline.
Global Motion Perception | Pre- and post-treatment (Days 1-5); 24-hour follow-up (Day 6); 72-hour follow-up (Day 8); and 10-day follow-up (Day 15).
  A change in global motion perception coherence threshold (%) from baseline.
Form Pattern Recognition | Pre- and post-treatment (Days 1-5); 24-hour follow-up (Day 6); 72-hour follow-up (Day 8); and 10-day follow-up (Day 15).
  A change in form pattern recognition coherence threshold (%) from baseline.
Pattern-reversal Visual Evoked Potentials (pVEP) | Pre-treatment (Day 1); post-treatment (Day 5); 24-hour follow-up (Day 6); 72-hour follow-up (Day 8); and 10-day follow-up (Day 15).
  A change in N75-P100 amplitudes and P100 latencies from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University Eye Institute, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding Z, Li J, Spiegel DP, Chen Z, Chan L, Luo G, Yuan J, Deng D, Yu M, Thompson B. The effect of transcranial direct current stimulation on contrast sensitivity and visual evoked potential amplitude in adults with amblyopia. Sci Rep. 2016 Jan 14;6:19280. doi: 10.1038/srep19280. PMID 26763954
- [Background] Thompson B, Mansouri B, Koski L, Hess RF. Brain plasticity in the adult: modulation of function in amblyopia with rTMS. Curr Biol. 2008 Jul 22;18(14):1067-71. doi: 10.1016/j.cub.2008.06.052. PMID 18635353
- [Background] Thompson B, Mansouri B, Koski L, Hess RF. From motor cortex to visual cortex: the application of noninvasive brain stimulation to amblyopia. Dev Psychobiol. 2012 Apr;54(3):263-73. doi: 10.1002/dev.20509. Epub 2010 Nov 8. PMID 22415915
- [Background] Clavagnier S, Thompson B, Hess RF. Long lasting effects of daily theta burst rTMS sessions in the human amblyopic cortex. Brain Stimul. 2013 Nov;6(6):860-7. doi: 10.1016/j.brs.2013.04.002. Epub 2013 Apr 28. PMID 23664756